CLINICAL TRIAL: NCT04121650
Title: Executive Functions and Symptom Reduction in Youth Receiving Home-based Treatment With Collaborative Problem Solving
Brief Title: Executive Function and Symptom Reduction in Youth Receiving Home-based Treatment With Collaborative Problem Solving
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Gerstner Philanthropies (Unknown); Youth Villages (Other)
Responsible Party: Principal Investigator, Alisha R Pollastri, Director of Research and Evaluation, Think:Kids, Massachusetts General Hospital
Other Study IDs: 2019P002239
Record Dates: First submitted 2019-10-07; First posted 2019-10-10 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Child Behavior; Problem Behavior; Executive Dysfunction
Keywords: Executive Functioning; ADHD; Behavior Problems; Youth; CPS; Collaborative Problem Solving; Disruptive Behavior; Parenting
MeSH Terms: conditions — Child Behavior; Problem Behavior; Attention Deficit Disorder with Hyperactivity; Mental Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Collaborative Problem Solving — CPS is an approach for understanding and reducing challenging behavior in youth. Under CPS, caregivers are taught to understand and identify the specific neurocognitive skill deficits that underlie their child's challenging behavior. Then the caregivers are taught to interact with the child in a way that solves chronic behavior problems while building the lagging neurocognitive skills to avoid future problems.
  Other Names: CPS

SUMMARY:
In this project, the investigators will extend prior results of parent-reported executive function growth and symptom reduction in children receiving home-based treatment with the Collaborative Problem Solving treatment approach (CPS), with a particular focus on examining children who have attention deficit hyperactivity disorder (ADHD). The investigators will examine executive functioning (EF) of children who are receiving CPS, measuring EF with parent-report and objective computer-based tasks, at two timepoints: at the start of treatment and approximately four months later, and will collect symptoms at these plus three additional timepoints: at discharge, 6-months after discharge, and 12-months after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Clients of participating non-profit organization that are receiving home-based youth mental health care
* Speaking and writing English at level necessary to complete study requirements

Exclusion Criteria:

* Youth is in full state custody and consent cannot be obtained by a guardian
* Youth and/or guardians do not speak English well enough to complete standardized measures
* Youth has a confirmed or suspected Full Scale IQ below 70, or carries a prior diagnosis of Autism Spectrum Disorder at the moderate or severe level

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The participants of this study are youth (ages 7 to 14) who are the identified clients being seen in home-based therapy at identified Youth Villages sites in Massachusetts.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in Behavioral Symptoms | Baseline, 4 months, discharge, 6 months post-discharge, and 12 months post-discharge
  Strengths and Difficulties Questionnaire (Parent-report measuring child emotional problems, conduct issues, hyperactivity/inattention, peer relationship problems, and pro- social behavior)
Change in Behavioral Symptoms | Baseline, 4 months, and discharge
  Clinical Global Impressions (Measures clients' symptom severity, global improvement, and therapeutic response)
Change in Executive Functioning Skills | Baseline and 4 months
  Behavior Rating Inventory of Executive Functioning (Parent-report measuring deficits in different domains of executive functioning)
Change in Executive Functioning Skills | Baseline and 4 months
  CANTAB computer-based cognitive tasks (Motor Screening Task, Stop Signal Task, Spatial Span, Multitasking Test, Stockings of Cambridge, Intra-Extra Dimensional Set Shift)

SECONDARY OUTCOMES:
Change in Child-Parent Relationship | Baseline and 4 months
  Child-Parent Relationship Scale (A 15-question measure of parents perceptions of their relationship with their child by using a scale of 1-5 where 1 "definitely does not apply" and a 5 "definitely applies to the child-parent relationship")
Treatment providers' fidelity to Collaborative Problem Solving (as a moderator) | provider rating made closest in proximity to four-month timepoint
  CPS Treatment Integrity Rating Form Short (Observational ratings by trained CPS coaches that quantitatively measure providers' fidelity to the practice of the CPS treatment approach)

CONTACTS AND LOCATIONS:
Overall Officials: Alisha R Pollastri, Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States